CLINICAL TRIAL: NCT05792072
Title: High Frequency rTMS for the Treatment of Neuropathic Pain in Diabetic Patients
Brief Title: rTMS for the Treatment of Neuropathic Pain in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMSDIAB2021
Record Dates: First submitted 2022-12-07; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-09

CONDITIONS: Neuropathic Pain; Diabetic Neuropathies
MeSH Terms: conditions — Neuralgia; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS (Active Comparator): The patient will receive one daily rTMS session for 5 days of HF-rTMS, delivered through an H-coil applied to the primary motor area of the leg. Each session will last 20 minutes during which 30 consecutive trains of 50 stimuli will be delivered at 20 Hz at 100% of resting motor threshold (RMT), with an intertrain interval of 30s
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): Sham stimulation will be delivered using a sham coil.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — High-frequency rTMS
  Arms: active rTMS
Device: Sham rTMS — sham rTMS
  Arms: Sham rTMS

SUMMARY:
Tis study aims to assess whether multiple sessions of sham-controlled HF-rTMS applied to the motor cortex significantly reduces treatment-resistant neuropathic pain in diabetic patients.

This study will also investigate the effect of those rTMS sessions on functional connectivity of the M1 with brain areas involved in pain processing, underlying brain metabolism and brain plasticity using rs-fMRI, MRS and Paired-pulse stimulation respectively in those patients.

Subjects will be randomized into two groups to receive real or sham rTMS protocol. A washout period of at least 8 weeks will be respected between protocols to minimize carry-over effects. Sham stimulation will be delivered using a sham coil, providing the same auditory and sensory stimuli.

One daily rTMS session for 5 days of HF-rTMS, will be delivered through an H-coil applied to the primary motor area of the leg. Each session will last 20 minutes during which 30 consecutive trains of 50 stimuli will be delivered at 20 Hz at 100% of resting motor threshold (RMT), with an intertrain interval of 30s

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this study is obtained
* The subject is an out-patient aged 18 years or above with diabetes mellitus type 1 or 2
* The patient has laboratory-confirmed diabetes
* Patients are diagnosed with peripheral neuropathy based on clinical and electrophysiological findings
* A score of > /= 4 on the the 'Douleur Neuropathique en 4 Questions' (DN4) questionnaire (30), conforming the diagnosis of neuropathic pain.
* The patient has a painful diabetic neuropathy for at least 6 months
* The patient has a Numeric pain rating scale (NPRS) score >/= 4.
* The patient is resistant to standard therapies for neuropathic pain

Exclusion Criteria:

* The patient has an implanted cardiac device, such as a pacemaker or a defibrillator
* The patient has an implanted neurostimulator
* The patient has cochlear implants/ear implants, magnetic dental im-plants
* The patient has a drug infusion pump
* The patient has cerebral artery aneurysm clips
* The patient has a history of epilepsy
* The patient has a history of migraine or severe headaches
* The patient has significant psychiatric disorders
* For female patients: the subject is pregnant or lactating
* Other formal contra-indication for rTMS or MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-02 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Changes in pain severity | The NPRS will be controlled at following time points: prior to the initiation of the rTMS protocol, and then weekly until 2 months after the last treatment.
  Neuropathic pain rating scale; Scores are based on patient responses to questions about pain intensity. 0 indicates no pain; 10 indicates the most pain imaginable
Changes in functional connectivity of the M1 with brain areas involved in pain processing | rs-fMRI will be controlled at baseline before active or sham rTMS, 1 week after active rTMS and sham rTMS, 2 weeks after active and sham rTMS, 2 months after the last treatment
  rs-fMRI will be used
Changes in brain metabolism | MRS will be controlled at baseline before active or sham rTMS, 1 week after active rTMS and sham rTMS, 2 weeks after active and sham rTMS, 2 months after the last treatment
  MRS will be used
Changes in brain plasticity | Paired-pulse stimulation will be controlled at baseline before active or sham rTMS, 1 week after active rTMS and sham rTMS, 2 weeks after active and sham rTMS, 2 months after the last treatment
  Paired-pulse stimulation will be used

SECONDARY OUTCOMES:
Influence on the quality of life | Will be controlled at baseline before active or sham rTMS, 1 week after active rTMS and sham rTMS, 2 weeks after active and sham rTMS, 2 months after the last treatment
  RAND 36-Item Health Survey; It is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions.
  Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. A high score defines a more favorable health state.
influence on depression | Will be controlled at baseline before active or sham rTMS, 1 week after active rTMS and sham rTMS, 2 weeks after active and sham rTMS, 2 months after the last treatment
  Beck Depression Inventory (BDI-II); total scores ranging from 0 to 63. Higher total scores indicate more severe depressive symptoms
influence on nerve conduction | this wil be controlled at baseline and 2 months after the last treatment.
  Electrodiagnostic testing: This involves nerve conduction studies (NCS) and electromyography (EMG) testing.
  During NCS the following measurements will be performed:
  * Motor conduction of the peroneal nerve, median motor study
  * sensory conduction of the sural nerves, median and ulnar nerve
  * Soleus H-reflex
  * Sympathic skin respons
  EMG study of distal and proximal muscles of at least one upper and lower extremity will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Brussels, Brussels, Jette, Belgium